CLINICAL TRIAL: NCT02096640
Title: Randomized Controlled Trial on the Effect of Percutaneous Dilatation Tracheostomy Compared to Open Surgical Tracheostomy on Postoperative Inflammation, Pulmonary Function, Peri- and Postoperative Complications and Physical Mobilization.
Brief Title: Postoperative Inflammation and Recovery After Tracheostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Markus Castegren, Med. dr., Sormland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1136-31/2; 2013/1136-31/2LTS (Other: Sormlands Landsting)
Record Dates: First submitted 2014-03-13; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Tracheostomy Complication; Inflammation; Post-operative Complications
MeSH Terms: conditions — Inflammation | interventions — Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous dilatation tracheostomy: Smiths Medical (Active Comparator): Type of surgical teqnique for tracheostomy: Percutaneous dilatation tracheostomy. The set for the tracheostomy is bought from Smiths Medical TM.
  Interventions: Procedure: Type of surgical teqnique for tracheostomy
- Open surgery tracheostomy (Active Comparator): Type of surgical teqnique for tracheostomy: Open surgical tracheostomy
  Interventions: Procedure: Type of surgical teqnique for tracheostomy

INTERVENTIONS:
Procedure: Type of surgical teqnique for tracheostomy

SUMMARY:
The main purpose of this study is to examine if there are differences in postoperative inflammation following percutaneous dilatation tracheostomy versus surgical tracheostomy in intensive care unit patients.

DETAILED DESCRIPTION:
Are there differences between the two arms in plasma concentrations of inflammatory mediators (TNF-alfa, interleukin 1, 6, 10) at 24 hrs following the start of the surgical procedure? Are there differences between the two arms in the incidence of postoperative complications (i.e. bleeding, incidence of stomal infections, tracheal tube dislocation, airway compromisation), postoperative pulmonary infection (during the stay in the ICU) and pulmonary function (FEV1, dynamic complicance, oxygen demand, time to weaning off the ventilator: all measured daily during the ICU-stay), postoperative mobilization (time to mobilization to sitting, standing and walking, respectively)?

ELIGIBILITY:
Inclusion Criteria: Patients in whom a tracheostomy is indicated (i.e. anticipated need of mechanical ventilation for >7 days or anticipated risk for complicated extubation, e.g. anatomical signs of a compromised airway, reduced level of consciousness. Adults over 18 years. Participants who are suitable for both surgery techniques.

Exclusion Criteria:

Children under 18 years, pregnancy and participants with anatomical defects that exclude them from percutaneous dilatation tracheostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in inflammation markers in plasma | Preoperative and 24 hours after the start of surgery
  Plasma samples will be taken preoperative and 24 hours after the start of tracheostomy. The levels of TNF-alpha, IL-6 and IL-10 will be measured.

SECONDARY OUTCOMES:
Postoperative complications | Until discharge from the ICU
  All postoperative complications will be noted daily during the ICU-stay, i.e. bleeding, incidence of stomal infections, tracheal tube dislocation, airway compromisation.

OTHER OUTCOMES:
Physical function | One week after tracheostomy
  Notes 7 Days after tracheostomy on the time to mobilization to sitting, standing and walking, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Castegren, MD, PhD, Principal Investigator — Centre for Clinical Research, Uppsala University
Locations (1):
- Intensivvårdsavdelningen på Mälarsjukhuset, Eskilstuna, Sörmland, Sweden